CLINICAL TRIAL: NCT04528992
Title: Effects of Blood Flow Restriction (BFR) Therapy on Early Anterior Cruciate Ligament (ACL) Graft Maturation
Brief Title: Effects of Blood Flow Restriction (BFR) Therapy on ACL Graft Maturation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: BFR Physical Therapy Protocol was not finalized and department had multiple similar studies.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Seth Sherman, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-56716
Record Dates: First submitted 2020-08-18; First posted 2020-08-27 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Knee Injuries; Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Knee Injuries; Anterior Cruciate Ligament Injuries | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical Therapy with BFR (Experimental): Participants will begin BFR therapy as early as 2 weeks after surgery. The initial 2 weeks after surgery, or prior to initiation of BFR will consist of the physical therapy following the surgeon's postoperative protocol.
  Interventions: Other: Blood Flow Restriction Therapy
- Physical Therapy without BFR (Active Comparator): Participants will undergo standard physical therapy following the surgeon's postoperative protocol.
  Interventions: Other: Standard Postoperative Physical Therapy

INTERVENTIONS:
Other: Blood Flow Restriction Therapy — BFR is a rehabilitation method that involves wearing a tight band around the exercising extremity to briefly limit blood flow while doing light weight exercises. The response is similar to heavy weight training or lifting but without the stress on the extremity that is still healing from surgery. Will be given after 2 weeks standard postoperative physical therapy per surgeon's ACL reconstruction protocol following surgery.
  Arms: Physical Therapy with BFR
Other: Standard Postoperative Physical Therapy — This is the surgeon's standard postoperative physical therapy protocol after ACL reconstruction.
  Arms: Physical Therapy without BFR

SUMMARY:
This is a study comparing the effects of blood flow restriction (BFR) therapy on the maturation of the Anterior Cruciate Ligament (ACL) graft after reconstruction surgery compared to physical therapy without the use of BFR.

DETAILED DESCRIPTION:
The study will be a randomized controlled trial to compare outcomes between physical therapy with BFR and physical therapy without BFR on the ACL graft maturation following reconstruction surgery. BFR therapy will begin as early as 2 weeks after surgery. The initial 2 weeks after surgery, or prior to initiation of BFR, will consist of the physical therapy following the surgeon's postoperative protocol.

To be considered for participation in this study, patients must be 18 years and older undergoing primary ACL reconstruction. In addition, patients must meet several inclusion/exclusion criteria to be randomized and included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 or older, all gender
* Patients receiving any type of ACL graft, either autograft or allograft, and any type of tissue

Exclusion Criteria:

* Patients who do not meet the the comprehensive BFR screening criteria based on predetermined contraindications and precautions
* Patients undergoing any additional concomitant ligament repair or reconstruction at the same surgery
* Revision procedures
* Patients unable to lay still in an MRI scanner
* Patients receiving treatment outside Stanford
* Patients undergoing concomitant meniscus treatment that restricts patients' weight bearing or prolongs their immobilization compared to their surgeons standard postoperative ACL reconstruction protocol
* Patients who are unable to lay still in an MRI scanner
* Patients with a torn ACL or previous ACL reconstruction in the contralateral knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Difference in MRI imaging of Graft | 2 weeks, 3 months, 6 months
  Graft ligamentization or maturation on MRI using T2 mapping
Difference in Quadriceps Volume & Cross-sectional Area | 3 months, 6 months
  Quadriceps muscle atrophy measured on MRI with quadriceps cross-sectional area
Difference in Thigh Circumference Measurement | 3 months, 6 months
  Muscle measurement determined with measuring tape for thigh circumference

SECONDARY OUTCOMES:
Isokinetic Dynamometer | 2 weeks, 3 months, 6 months
  Measurement of knee extension and flexion torque at 180° and 300°/sec using the isokinetic dynamometer
Visual Analog Scale (VAS) | 2 weeks, 3 months, 6 months
  Patient reported assessment of current level of pain from no pain to worst imaginable
Single Assessment Numerical Evaluation (SANE) | 2 weeks, 3 months, 6 months
  Patient reported outcome measure of function. 0-100% scale with 100% being normal
International Knee Documentation Committee (IKDC) | 2 weeks, 3 months, 6 months
  Patient reported outcome measure of symptoms, sports activity & knee function. 0-100 points with 0 (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Seth Sherman, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford, Redwood City, California, United States